CLINICAL TRIAL: NCT04185402
Title: Azithromycin Reduction to Reach Elimination of Trachoma
Acronym: ARRET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Programme National de Santé Oculaire (PNSO) (Unknown); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-28923; 5UG1EY030833 (NIH)
Record Dates: First submitted 2019-12-02; First posted 2019-12-04 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Trachoma
MeSH Terms: conditions — Trachoma | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Azithromycin Continuation (Active Comparator): In study communities randomized to the Azithromycin Continuation arm, all individuals aged 1 month and older will receive a single mass distribution of azithromycin several weeks after the baseline and 36-month monitoring visits. Oral azithromycin, 20 mg/kg for children and 1 g for adults, will be offered to all households identified on the preceding census in the communities randomized to continuing treatment. Study drug will be distributed by health extension workers and organized by PNSO. Individuals with a known macrolide allergy will be offered a two-week course of daily ophthalmic tetracycline ointment (two tubes).
  Interventions: Drug: Azithromycin
- Azithromycin Discontinuation (No Intervention): In study communities randomized to the Azithromycin Discontinuation arm, individuals will receive no treatment.

INTERVENTIONS:
Drug: Azithromycin — In study communities randomized to the Azithromycin Continuation arm, all individuals aged 1 month and older will receive a single mass distribution of azithromycin several weeks after the baseline and 36-month monitoring visits. In study communities randomized to Azithromycin Discontinuation, participants will receive no treatment.
  Arms: Azithromycin Continuation

SUMMARY:
The investigators propose a randomized controlled trial of discontinuation versus continuation of annual mass azithromycin distribution in hypoendemic communities of Maradi, Niger. The investigators will randomize communities with up to 20% Trachomatous Inflammation - Follicular (TF) prevalence following at least 5 years of mass azithromycin distribution to discontinuation or continuation of 3 additional years of annual mass azithromycin distribution.

ELIGIBILITY:
Inclusion Criteria:

* Provision of appropriate informed consent
* Stated willingness to comply with all study procedures
* Live in one of the 80 communities with up to 20% prevalence of TF selected for the trial

Exclusion Criteria:

* Does not consent to participation
* Unwilling to comply with all study procedures
* Does not live in one of the 80 communities with up to 20% prevalence of TF selected for the trial

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 74920 (Actual)
Dates: Start 2021-05-29 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Ocular chlamydia measured in a population-based sample of 0-9 year-old children | 36 months
  Assessed by PCR

SECONDARY OUTCOMES:
Infectious load of chlamydia among 0-9 year-old children infected with ocular chlamydia | 36 months
  Assessed by PCR
Conjunctival inflammation | 36 months
  Assessed from conjunctival photography. Clinical photographs of the conjunctiva will be assessed by masked graders according to the grading scale described by the WHO Simplified Grading System.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Oldenburg, ScD, MPH, Principal Investigator — University of California, San Francisco; Tom Lietman, MD, Principal Investigator — University of California, San Francisco; Elodie Lebas, RN, Study Director — University of California, San Francisco
Locations (1):
- Programme National de Santé Oculaire (PNSO), Niamey, Niger

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amza A, Kadri B, Nassirou B, Arzika AM, Austin A, Nyatigo F, Lebas E, Arnold BF, Lietman TM, Oldenburg CE. Azithromycin Reduction to Reach Elimination of Trachoma (ARRET): study protocol for a cluster randomized trial of stopping mass azithromycin distribution for trachoma. BMC Ophthalmol. 2021 Jan 6;21(1):15. doi: 10.1186/s12886-020-01776-4. PMID 33407263